CLINICAL TRIAL: NCT02881398
Title: A Randomized Trial of Pocket-Echocardiography Integrated Mobile Health Device Assessments in Modern Structural Heart Disease Clinics
Brief Title: Mobile Health in Structural Heart Disease
Acronym: ASEF-VALUES
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sri Sathya Sai Institute of Higher Medical Sciences (Other)
Responsible Party: Principal Investigator, Srikanth Sola, Additional Senior Consultant, Sri Sathya Sai Institute of Higher Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ASEF-VALUES
Record Dates: First submitted 2016-08-18; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatic Heart Disease; Heart Diseases
Keywords: Mobile Health; Telemedicine; Pocket-Echocardiography
MeSH Terms: conditions — Rheumatic Heart Disease; Heart Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mHealth (Experimental): Each participant randomized to a mHealth assessment were evaluated with: (1) structural abnormalities with handheld-echocardiography (Vscan®, General Electric Healthcare); (2) vital signs with smartphone-connected oxymetry and blood pressure monitors (iHealthLabs®); (3) functional assessments on a 6-minute walk test with a trial-axial activity monitor (Ozeri®); (4) cardiac rhythm abnormalities with smartphone-connected- iECG (AliveCor®) and; (5)point-of-care testing with fingerstick B-type natriuretic peptide (Alere). All study participants then underwent a comprehensive transthoracic echocardiogram for anatomical assessments of the severity of rheumatic and structural heart disease prior to percutaneous valvuloplasty or a surgical valve replacement.
  Interventions: Device: mHealth
- Standard-Care (Active Comparator): Each participant randomized to a standard-assessment were evaluated with the resource available at the institution including a physical examination,12 lead-ECG, radiographic, laboratory testing as clinically required. All study participants underwent a comprehensive transthoracic echocardiogram for anatomical assessments of the severity of rheumatic and structural heart disease prior to percutaneous valvuloplasty or a surgical valve replacement.
  Interventions: Other: Standard-Care

INTERVENTIONS:
Device: mHealth — After randomization and at the time of the initial encounter, study subjects are assessed at the point-of-care with mHealth devices that measure symptoms, functional status, and for structural abnormalities. These devices include activity monitoring for an assessment of a 6-minute walk test, smartphone connected blood pressure, oxymetry and ECG for functional assessments, and structural assessments with handheld-echocardiography and point-of-care BNP. Treatment decisions for an intervention with percutaneous valvuloplasty or valve replacement were performed based on the aggregate of these mHealth findings. Confirmation of the severity of structural heart disease on transthoracic echocardiography was performed on all participants.
  Arms: mHealth
Other: Standard-Care — After randomization and at the time of the initial encounter, study subjects randomized to standard-care underwent a physical examination, 12-lead ECG, radiographic and laboratory tests as warranted and clinically required. Treatment decisions for percutaneous valvuloplasty or valve replacement were based on the aggregate of the standard-care findings. Confirmation of the severity of structural heart disease on transthoracic echocardiography was performed on all participants.
  Arms: Standard-Care

SUMMARY:
The primary objective of this investigation was to assess the impact of new mobile health devices on health outcomes among patients with rheumatic and structural heart disease in a resource limited area. To achieve this aim the investigators utilized smartphone-connected devices such as the smartphone-ECG, activity monitors, connected blood pressure devices and pocket-sized and handheld ultrasound. The main question asked in this investigation is if mobile health assessments accelerates medical-decision-making and if it shortens the time to definitive therapy.

DETAILED DESCRIPTION:
A recent paradigm-shift in the global burden of cardiovascular diseases has been observed with a decreasing prevalence in industrialized nations and an increasing prevalence in resource limited areas. This problem is further compounded with resource-limited areas receiving a disproportionately low allocation of global resources including diagnostic tests and trained healthcare professionals. Such cardiovascular conditions include heart failure, coronary artery disease, atrial arrhythmias and hypertensive heart disease. Coupled with a rising epidemic of rheumatic and structural heart disease affecting over 15- million individuals in these regions creates an urgent need that requires innovative and scalable methods to improve population- health, methods that reduce the cost of care, and simultaneously improves outcomes.

The World Health Organization's Millennium Developmental Goals has recently reported a rise in cellular phone technologies with 7-Billion devices in active circulation. Parallel developments with the globalization of Internet-based communication and the emergence of new smartphone-connected mobile health (mHealth) devices are providing new methods for patients to remotely monitor their chronic conditions and for providers to improve healthcare delivery. These technologies include smartphone 'apps', wearable and wireless devices such as the smartphone-ECG, sensor-based technologies, pocket-sized ultrasound and miniaturized lab-on-a-chip technologies. Several design features of mHealth are well suited for use in resource-limited areas and used as a practitioner-based diagnostic tool including portability, lower cost, and simple to use form factors. Although an attractive method for new technology utilization, the impact of mHealth used as a practitioner-based clinical-decision-support tool on subsequent management and outcomes has not been previously evaluated.

Several barriers to effective healthcare exist in resource-limited areas that requires multidisciplinary collaborations between the community, medical centers, health workers and patients. Developing new digital programs with healthcare innovations in these regions brings together a collaboration of industry, researchers, engineers and information technology partners. In the aggregate, a cumulative effort across several disciplines is necessary in order to assess the feasibility, utility, and impact of new devices in resource constrained areas. The investigators describe a multidisciplinary and global effort across institutions in India and the United States. The investigators received support from international medical societies and device manufacturers to advance our knowledge for technology utilization and to improve healthcare access and outcomes for patients in resource limited areas.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic outpatients with a new or an established diagnosis of rheumatic and structural heart disease and included valvular disease, left/right ventricular failure, rheumatic valvular disease, congenital heart defects and included adult, pediatric, and pregnant patients. Patients with a prior valvuloplasty or valve replacement for structural heart disease were also included

Exclusion Criteria:

* Exclusions included neonatal patients and those with an unstable hemodynamic status

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Time to definitive treatment with Valvuloplasty or Valve Replacement | Upto 12 months after enrollment

SECONDARY OUTCOMES:
Cardiovascular Hospitalization and/or Death | Upto 12 months after enrollment
  Secondary outcomes included the occurrence of a cardiovascular hospitalization and/or death over 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Srikanth Sola, MD, Principal Investigator — Sri Sathya Sai Institute of Higher Medical Sciences; Sanjeev Bhavnani, MD, Study Director — Scripps Clinic and Reseach Institute; Partho Sengupta, MD, Principal Investigator — Icahn School of Medicine at Mt. Sinai

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to requesting investigators and 6 months after publication

REFERENCES:
- [Background] Singh S, Bansal M, Maheshwari P, Adams D, Sengupta SP, Price R, Dantin L, Smith M, Kasliwal RR, Pellikka PA, Thomas JD, Narula J, Sengupta PP; ASE-REWARD Study Investigators. American Society of Echocardiography: Remote Echocardiography with Web-Based Assessments for Referrals at a Distance (ASE-REWARD) Study. J Am Soc Echocardiogr. 2013 Mar;26(3):221-33. doi: 10.1016/j.echo.2012.12.012. PMID 23439071
- [Background] Bansal M, Singh S, Maheshwari P, Adams D, McCulloch ML, Dada T, Sengupta SP, Kasliwal RR, Pellikka PA, Sengupta PP; VISION-in-Tele-Echo Study Investigators. Value of interactive scanning for improving the outcome of new-learners in transcontinental tele-echocardiography (VISION-in-Tele-Echo) study. J Am Soc Echocardiogr. 2015 Jan;28(1):75-87. doi: 10.1016/j.echo.2014.09.001. Epub 2014 Oct 8. PMID 25306222
- [Background] Bhavnani SP, Narula J, Sengupta PP. Mobile technology and the digitization of healthcare. Eur Heart J. 2016 May 7;37(18):1428-38. doi: 10.1093/eurheartj/ehv770. Epub 2016 Feb 11. PMID 26873093
- [Background] Bansal M, Sengupta PP. Setting global standards in adult echocardiography: Where are we? Indian Heart J. 2015 Jul-Aug;67(4):298-301. doi: 10.1016/j.ihj.2015.07.020. Epub 2015 Aug 21. No abstract available. PMID 26304560
- [Background] Drain PK, Hyle EP, Noubary F, Freedberg KA, Wilson D, Bishai WR, Rodriguez W, Bassett IV. Diagnostic point-of-care tests in resource-limited settings. Lancet Infect Dis. 2014 Mar;14(3):239-49. doi: 10.1016/S1473-3099(13)70250-0. Epub 2013 Dec 10. PMID 24332389
- [Background] Yusuf S, Rangarajan S, Teo K, Islam S, Li W, Liu L, Bo J, Lou Q, Lu F, Liu T, Yu L, Zhang S, Mony P, Swaminathan S, Mohan V, Gupta R, Kumar R, Vijayakumar K, Lear S, Anand S, Wielgosz A, Diaz R, Avezum A, Lopez-Jaramillo P, Lanas F, Yusoff K, Ismail N, Iqbal R, Rahman O, Rosengren A, Yusufali A, Kelishadi R, Kruger A, Puoane T, Szuba A, Chifamba J, Oguz A, McQueen M, McKee M, Dagenais G; PURE Investigators. Cardiovascular risk and events in 17 low-, middle-, and high-income countries. N Engl J Med. 2014 Aug 28;371(9):818-27. doi: 10.1056/NEJMoa1311890. PMID 25162888
- [Background] Marijon E, Ou P, Celermajer DS, Ferreira B, Mocumbi AO, Jani D, Paquet C, Jacob S, Sidi D, Jouven X. Prevalence of rheumatic heart disease detected by echocardiographic screening. N Engl J Med. 2007 Aug 2;357(5):470-6. doi: 10.1056/NEJMoa065085. PMID 17671255
- [Background] Engelman D, Kado JH, Remenyi B, Colquhoun SM, Carapetis JR, Donath S, Wilson NJ, Steer AC. Focused cardiac ultrasound screening for rheumatic heart disease by briefly trained health workers: a study of diagnostic accuracy. Lancet Glob Health. 2016 Jun;4(6):e386-94. doi: 10.1016/S2214-109X(16)30065-1. PMID 27198843
- [Background] Mirabel M, Bacquelin R, Tafflet M, Robillard C, Huon B, Corsenac P, de Fremicourt I, Narayanan K, Meunier JM, Noel B, Hagege AA, Rouchon B, Jouven X, Marijon E. Screening for rheumatic heart disease: evaluation of a focused cardiac ultrasound approach. Circ Cardiovasc Imaging. 2015 Jan;8(1):e002324. doi: 10.1161/CIRCIMAGING.114.002324. PMID 25567654
- [Derived] Bhavnani SP, Sola S, Adams D, Venkateshvaran A, Dash PK, Sengupta PP; ASEF-VALUES Investigators. A Randomized Trial of Pocket-Echocardiography Integrated Mobile Health Device Assessments in Modern Structural Heart Disease Clinics. JACC Cardiovasc Imaging. 2018 Apr;11(4):546-557. doi: 10.1016/j.jcmg.2017.06.019. Epub 2017 Oct 5. PMID 28917688